CLINICAL TRIAL: NCT05680233
Title: A Phase 1a/1b Single Ascending and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of OA-235i, a PAR2 Inhibitor, in Adults With Nonalcoholic Steatohepatitis
Brief Title: Safety Study of OA-235i in Subjects With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oasis Pharmaceuticals, LLC (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OAS-235i-101; 5R44DK101240 (NIH)
Record Dates: First submitted 2022-12-12; First posted 2023-01-11 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Nonalcoholic Steatohepatitis; Nonalcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Single ascending dose (SAD) sequential group study of a sc dose of OA-235i in five (5) planned dose cohorts with 3 subjects/cohort administering a bolus injection at escalating dose levels from 4 to 40 mg. One (1) planned multiple dose (MD), randomized, placebo-controlled expansion cohort with 9 NAFLD/NASH subjects will be enrolled for a 7-day dosing regimen at a dose level to be determined from the SAD portion of the study.
Masking Description: All subjects will be blinded to IP dose/level in Phase 1a; subjects, Investigator and site staff (excluding unblinded pharmacy staff) will be blinded to IP/placebo in Phase 1b.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OA-235i (4-40 mg) (Experimental): Single ascending dose (SAD): OA-235i (4-40 mg) administered subcutaneously (SC) once to adult subjects with suspected or confirmed diagnosis of noncirrhotic nonalcoholic fatty liver disease (NAFLD)/nonalcoholic steatohepatitis (NASH) without advanced hepatic fibrosis.
  Multiple dose (MD): OA-235i (dose level to be determined from SAD) or placebo administered subcutaneously (SC) once daily for 7 days to adult subjects with suspected or confirmed diagnosis of noncirrhotic nonalcoholic fatty liver disease (NAFLD)/nonalcoholic steatohepatitis (NASH) without advanced hepatic fibrosis.
  Interventions: Drug: OA-235i (4 mg); Drug: OA-235i (8 mg); Drug: OA-235i (16 mg); Drug: OA-235i (30 mg); Drug: OA-235i (40 mg); Drug: OA-235i or placebo

INTERVENTIONS:
Drug: OA-235i (4 mg) — 3 participants will receive 4 mg as a single subcutaneous dose
  Other Names: PAR2 inhibitor
Drug: OA-235i (8 mg) — 3 participants will receive 8 mg as a single subcutaneous dose
  Other Names: PAR2 inhibitor
Drug: OA-235i (16 mg) — 3 participants will receive 16 mg as a single subcutaneous dose
  Other Names: PAR2 inhibitor
Drug: OA-235i (30 mg) — 3 participants will receive 30 mg as a single subcutaneous dose
  Other Names: PAR2 inhibitor
Drug: OA-235i (40 mg) — 3 participants will receive 40 mg as a single subcutaneous dose
  Other Names: PAR2 inhibitor
Drug: OA-235i or placebo — 9 participants will receive a daily subcutaneous dose of OA-235i or placebo for 7 consecutive days
  Other Names: PAR2 inhibitor; placebo

SUMMARY:
This study is a Phase 1, first-in-human single-dose escalation and multiple dose study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of OA-235i in subjects with nonalcoholic steatohepatitis.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single ascending dose (SAD) in participants with suspected or confirmed diagnosis of noncirrhotic nonalcoholic fatty liver disease (NAFLD)/nonalcoholic steatohepatitis (NASH) without advanced hepatic fibrosis. This dose-escalating strategy will test the safety of OA-235i when given as a single subcutaneous dosage using up to five successive cohorts. Each cohort will have three non-randomized participants receiving the active medication. One (1) planned multiple dose (MD) randomized, placebo-controlled expansion cohort with 9 NAFLD/NASH subjects will be enrolled for a 7-day dosing regimen at a dose level to be determined from the SAD portion of the study.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male and female subjects between the ages of 18 and 70 years, inclusive, at Screening.
2. Suspected or confirmed diagnosis of noncirrhotic NAFLD/NASH without advanced hepatic fibrosis by one of the following:

   1. Histologically with liver biopsy within 2 years prior to Screening (documentation with pathology report); or
   2. Radiologically with ≥5% steatosis measured by magnetic resonance imaging-derived proton density fat fraction (MRI-PDFF), or controlled attenuation parameter (CAP) >238 dB/m via FibroScan assessment, or presence of hepatic steatosis on abdominal ultrasound ; or
   3. Clinically with a diagnosis of Metabolic Syndrome (MetS) reflecting the presence of at least 3 of 5 factors/criteria (ie, abdominal obesity, elevated triglycerides, reduced HDL-C, elevated blood pressure, and/or elevated fasting glucose [IFG or type 2 diabetes mellitus]) as defined by the National Cholesterol Education Program's Adult Treatment Panel III (NCEP ATP III) [Grundy 2005]; and fatty liver on imaging within 1 year prior to Screening.

Key Exclusion Criteria:

1. History or presence of cirrhosis as assessed by Investigator following review of diagnostic measures (clinical, imaging, histopathology, or laboratory).
2. Clinical evidence of hepatic decompensation (laboratory or clinical abnormalities- ascites, variceal bleeding, etc.).
3. History or presence of other concomitant liver disease (eg, hepatitis B & C, alcoholic liver disease, autoimmune liver disease, primary biliary cirrhosis, primary sclerosing cholangitis, hemochromatosis, Wilson's disease, alpha-1 antitrypsin (A1AT) deficiency, bile duct obstruction, liver primary or metastatic cancer, drug-induced liver disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 30 Days
  Number of participants with treatment-emergent with adverse events (incidence and severity)

SECONDARY OUTCOMES:
To characterize the OA-235i Pharmacokinetics (PK) by Cmax | 8 Days
  OA-235i PK by peak plasma concentration (Cmax)
To characterize the OA-235i Pharmacokinetics (PK) by t1/2 | 8 Days
  OA-235i PK by the terminal elimination half-life (t1/2)
To characterize the OA-235i Pharmacokinetics (PK) by Tmax | 8 Days
  OA-235i PK by time to peak plasma concentration (Tmax)
To characterize the OA-235i Pharmacokinetics (PK) by AUC | 8 Days
  OA-235i PK by area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Athan Kuliopulos, MD, PhD, Study Director — Oasis Pharmaceuticals, LLC
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States